CLINICAL TRIAL: NCT01104155
Title: The Purpose of This Study is to Investigate Two Different Dose Regimens of Eribulin Mesylate in Combination With Intermittent Erlotinib in Patients With Previously Treated, Advanced Non-small Cell Lung Cancer
Brief Title: Eribulin Mesylate in Combination With Intermittent Erlotinib in Patients With Previously Treated, Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-G000-205
Record Dates: First submitted 2010-04-12; First posted 2010-04-15 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2018-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Eribulin Mesylate; Erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — eribulin; Erlotinib Hydrochloride

ARMS (2):
- eribulin mesylate, 21 day cycle (Active Comparator)
  Interventions: Drug: eribulin mesylate + erlotinib
- eribulin mesylate, 28 day cycle (Active Comparator)
  Interventions: Drug: eribulin mesylate + erlotinib

INTERVENTIONS:
Drug: eribulin mesylate + erlotinib — 21-day Regimen: Eribulin mesylate given at a dose of 2 mg/m2 as a 2-5 min intravenous (IV) bolus on Day 1 and 150 mg of erlotinib given orally once daily, one hour before or two hours after the ingestion of food, on Days 2-16 of a 21-day cycle.
  Arms: eribulin mesylate, 21 day cycle
Drug: eribulin mesylate + erlotinib — 28-day Regimen: Eribulin mesylate given at a dose of 1.4 mg/m2 as a 2-5 min IV bolus on Days 1 and 8, and 150 mg of erlotinib given orally once daily, one hour before or two hours after the ingestion of food, on Days 15-28 of a 28-day cycle.
  Arms: eribulin mesylate, 28 day cycle

SUMMARY:
This is a Phase 2, multicenter, randomized study of two different dose regimens of eribulin mesylate in combination with intermittent erlotinib in patients with previously treated, advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed non-small cell lung cancer (NSCLC)
* At least one prior platinum-based doublet anti-cancer treatment for recurrent or advanced NSCLC
* Disease progression during or after the last anti-cancer therapy
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Serum creatinine less than or equal to 2.0 mg/dL or creatinine clearance 40 mL/min according to Cockcroft and Gault formula:
* Absolute neutrophil count greater than or equal to 1.5 x 10^9/L, hemoglobin greater than or equal to 10 g/dL (can be corrected by growth factor or transfusion), and platelet count greater than or equal to 100 x 10^9/L
* Total bilirubin less than or equal to 1.5 times the upper limit of normal (ULN) and alkaline phosphatase (AP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 times ULN (in the case of liver metastases less than or equal to 5 times ULN). In case AP is greater than 3 times ULN (in absence of liver metastases) or greater than 5 times ULN (in presence of liver metastases) AND subject also is known to have bone metastases, the liver specific AP must be separated from the total and used to assess the liver function instead of the total AP.
* At least one lesion of greater than or equal to 1.5 cm in longest diameter for non-lymph nodes or greater than or equal to 1.5 cm in shortest diameter for lymph nodes which is serially measurable according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.17

  * Males and females, age greater than or equal to 18 years
  * Provide written informed consent
  * Are willing and able to comply with all aspects of the protocol
  * Females of childbearing potential must have a negative serum beta-human chorionic gonadotropin (Beta-hCG) at Visit 1 (Screening) and a negative urine pregnancy test prior to starting study drug (Visit 2). Female subjects of childbearing potential must agree to be abstinent or to use highly effective methods of contraception (eg, condom + spermicide, condom + diaphragm with spermicide, intrauterine device (IUD), or have a vasectomised partner) having starting for at least one menstrual cycle prior to starting study drugs and throughout the entire study period and for 30 days (longer if appropriate) after the last dose of study drug. Those women using hormonal contraceptives must also be using an additional approved method of contraception (as described previously). Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Male subjects who are not abstinent or have not undergone a successful vasectomy, who are partners of women of childbearing potential must use, or their partners must use a highly effective method of contraception (eg, condom + spermicide, condom + diaphragm with spermicide, IUD) starting for at least one menstrual cycle prior to starting study drugs and throughout the entire study period and for 30 days (longer if appropriate) after the last dose of study drug. Those with partners using hormonal contraceptives must also be using an additional approved method of contraception (as described previously).

Exclusion criteria:

* Prior therapy with eribulin or an tyrosine kinase inhibitor of the epidermal growth factor receptor
* Subjects with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued steroids for this indication for greater than or equal to 4 weeks before starting study treatment. Symptoms attributed to brain metastases must be stable for greater than or equal to 4 weeks before starting study treatment; radiographic stability should be determined by comparing contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI) brain scan performed during screening to a prior scan performed 4 weeks earlier.
* Existing anti-cancer therapy-related toxicities of grade greater than or equal to 2, other than any grade of alopecia or grade less than or equal to 2 neuropathy, which are acceptable
* Current smokers who will not stop smoking one week prior to treatment and during the study
* History of congestive heart failure with New York Heart Association (NYHA) Grade greater than II, unstable angina, myocardial infarction within the past 6 months, serious cardiac arrhythmia
* Electrocardiogram with QTc interval greater than or equal to 500 msec based upon Bazett's formula (QTcB)
* Females who are pregnant (positive Beta-hCG test) or breastfeeding
* Subject with hypersensitivity to eribulin and /or erlotinib or any of the excipients
* Presence of a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors
* Subjects who are known to be human immunodeficiency virus (HIV) positive, because the neutropenia caused by the study treatments may make such subjects particularly susceptible to infection
* Subjects with active viral hepatitis (A, B, or C) as demonstrated by positive serology
* Radiotherapy, chemotherapy, biological therapy or investigational agents within 2 weeks prior to start of study treatment
* Meningeal carcinomatosis
* History of drug or alcohol dependency or abuse within approximately the last 2 years
* Medically unfit to receive the study drug or unsuitable for any other reason according to investigator judgment
* Any history of or concomitant medical condition that, in the opinion of the Investigator, would compromise the subject's ability to safely complete the study
* Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-02-22 (Actual); Primary Completion 2011-04-07 (Actual); Study Completion 2017-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (64):
- United States (50):
  - Bessemer, Alabama
  - Birmingham, Alabama
  - Beverly Hills, California
  - La Jolla, California
  - Aurora, Colorado
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Lakewood, Colorado
  - Littleton, Colorado
  - Lone Tree, Colorado
  - Longmont, Colorado
  - Parker, Colorado
  - Thornton, Colorado
  - Washington D.C., District of Columbia
  - Ocala, Florida
  - Port Saint Lucie, Florida
  - Kansas City, Kansas
  - Overland Park, Kansas
  - Shawnee Mission, Kansas
  - Detroit, Michigan
  - Columbia, Missouri
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - Lee's Summit, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Elizabeth City, North Carolina
  - Portland, Oregon
  - Tualatin, Oregon
  - Philadelphia, Pennsylvania
  - East Providence, Rhode Island
  - Dallas, Texas
  - Fort Worth, Texas
  - Garland, Texas
  - Plano, Texas
  - Arlington, Virginia
  - Chesapeake, Virginia
  - Fairfax, Virginia
  - Gainesville, Virginia
  - Hampton, Virginia
  - Leesburg, Virginia
  - Newport News, Virginia
  - Norfolk, Virginia
  - Virginia Beach, Virginia
  - Williamsburg, Virginia
  - Winchester, Virginia
  - Woodbridge, Virginia
  - Spokane, Washington
  - Vancouver, Washington
- Hong Kong, Hong Kong
- Malaysia (2):
  - Kuantan, Pahang
  - George Town
- Singapore, Singapore
- South Korea (3):
  - Goyang
  - Gyeonggi-do
  - Seoul
- Taiwan (3):
  - Taichung
  - Tainan
  - Taipei
- Thailand (4):
  - Bangkok
  - Chiang Mai
  - Lampang
  - Songkhla

REFERENCES:
- [Derived] Mok TS, Geater SL, Iannotti N, Thongprasert S, Spira A, Smith D, Lee V, Lim WT, Reyderman L, Wang B, Gopalakrishna P, Garzon F, Xu L, Reynolds C. Randomized phase II study of two intercalated combinations of eribulin mesylate and erlotinib in patients with previously treated advanced non-small-cell lung cancer. Ann Oncol. 2014 Aug;25(8):1578-84. doi: 10.1093/annonc/mdu174. Epub 2014 May 14. PMID 24827127

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 164 participants were screened. Of these 164 participants, 41 were screening failures, and 123 were randomized into the study. Of the 41 screen failures, 31 participants failed to meet inclusion or exclusion criteria and 10 were excluded due to adverse events, withdrew consent, and other reasons.
Groups:
- Eribulin Mesylate Plus Erlotinib, 21 Day Regimen: Eribulin mesylate was given at a dose of 2 mg/m^2 as a 2 to 5 min intravenous (IV) bolus on Day 1 and 150 mg of erlotinib was given orally once daily, one hour before or two hours after the ingestion of food, on Days 2 to 16 of a 21-day cycle.
- Eribulin Mesylate Plus Erlotinib, 28 Day Regimen: Eribulin mesylate was given at a dose of 1.4 mg/m^2 as a 2 to 5 min IV bolus on Days 1 and 8, and 150 mg of erlotinib given orally once daily, one hour before or two hours after the ingestion of food, on Days 15 to 28 of a 28-day cycle.
Period: Overall Study
Arm/Group | Eribulin Mesylate Plus Erlotinib, 21 Day Regimen | Eribulin Mesylate Plus Erlotinib, 28 Day Regimen
Started | 63 | 60
Completed | 38 | 42
Not Completed | 25 | 18
Not completed — Adverse Event | 15 | 8
Not completed — Participant choice | 6 | 5
Not completed — Withdrawal of consent | 1 | 1
Not completed — Other | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eribulin Mesylate Plus Erlotinib, 21 Day Regimen | Eribulin Mesylate Plus Erlotinib, 28 Day Regimen | Total
Number analyzed (Participants) | 63 | 60 | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (11.08) | 63.1 (10.05) | 62.4 (10.57)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 33 | 33 | 66
  Gender: Female | 30 | 27 | 57

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants whose best overall response (BOR) was either a confirmed complete response (CR) or a partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria for target lesions assessed by computed tomography (CT) or magnetic resonance imaging (MRI) and based on investigator assessment. CRs and PRs had to be confirmed by a repeat assessment of response (CR or PR) separated by at least 4 weeks (28 days). CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to have a reduction in short axis to less than 10 millimeters. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR and the corresponding 95% two-sided confidence intervals (CI) were estimated for each treatment regimen using the Clopper-Pearson method for calculating the exact binomial CI. (CR + PR)
Time Frame: From date of first dose of study drug until, or up to the date of data cutoff (07 Apr 2011)
Population: Full analysis set (FAS) (Intent-to-treat population) included all participants who took at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eribulin Mesylate Plus Erlotinib, 21 Day Regimen | Eribulin Mesylate Plus Erlotinib, 28 Day Regimen
Number analyzed (Participants) | 63 | 60
Percentage of participants | 12.7 [5.6 to 23.5] | 16.7 [8.3 to 28.5]
Statistical Analysis 1: Comparison: Eribulin Mesylate Plus Erlotinib, 21 Day Regimen; Test type: Superiority or Other; p = 0.204, 1-sided exact binomial; Based on a one-sided exact binomial test compared to 9%
Statistical Analysis 2: Comparison: Eribulin Mesylate Plus Erlotinib, 28 Day Regimen; Test type: Superiority or Other; p = 0.041, 1-sided exact binomial

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR was assessed for participants with a BOR of CR or PR, and was defined as the time from first documented evidence of CR or PR (whichever status was recorded first) until the first documented sign of disease progression or death (due to any cause), whichever was first. DOR was defined for participants with a confirmed CR or PR. For participants in the subset of responders who did not progress or die, duration of response was censored. DOR was analyzed using the Kaplan-Meier method.
Time Frame: From date of first document CR or PR (whichever was recorded first) until first documentation of disease progression or death due to any cause, or up to data cutoff (31 May 2013) up to 3.25 years
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eribulin Mesylate Plus Erlotinib, 21 Day Regimen | Eribulin Mesylate Plus Erlotinib, 28 Day Regimen
Number analyzed (Participants) | 63 | 60
Months | 9.4 [2.7 to NA] — Not evaluable | 9.7 [5.6 to NA] — Not evaluable

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was measured as the time from the date of first administration of study treatment until the first documentation of disease progression or death (due to any cause), whichever occurred first, as determined by investigator assessment based on RECIST v1.1. Disease progression per RECIST v1.1 was defined as at least a 20% relative increase and 5 mm absolute increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. For participants who did not have an event (i.e. those who had not progressed, and were alive at the date of data cut-off or lost to Follow-up), progression-free survival was censored. Participants who did not progress in their disease were censored on the date of their last tumor assessment preceding the start of any additional anticancer therapy. PFS was analyzed using the Kaplan-Meier method.
Time Frame: From date of first dose of study drug until documentation of disease progression or death from any cause (whichever occurred first), or up to data cutoff (31 May 2013) up to 3.25 years
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eribulin Mesylate Plus Erlotinib, 21 Day Regimen | Eribulin Mesylate Plus Erlotinib, 28 Day Regimen
Number analyzed (Participants) | 63 | 60
Months | 3.5 [1.9 to 4.7] | 3.8 [3.3 to 5.5]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who had a BOR of CR or PR, or stable disease (SD; duration of SD lasted for at least 7 weeks). To be assigned a BOR of SD, the time from the first administration of study drug until the date of documented SD was to be greater than or equal to 7 weeks (49 days). A participant's tumor assessment had to be at least 7 weeks following the randomization date to be consider SD. DCR and the corresponding exact Clopper-Pearson 95% CI were computed by treatment regimen. (CR + PR + SD)
Time Frame: From date of first dose of study drug until documentation of disease progression or death from any cause (whichever occurred first) or up to data cutoff (31 May 2013), up to approximately 3.25 years
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eribulin Mesylate Plus Erlotinib, 21 Day Regimen | Eribulin Mesylate Plus Erlotinib, 28 Day Regimen
Number analyzed (Participants) | 63 | 60
Percentage of participants | 47.6 [34.9 to 60.6] | 63.3 [49.9 to 75.4]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the length of time in months from the date of first administration of study drug until the date of death from any cause, and was based on the data cutoff date. In the absence of confirmation of death, participants were censored either at the date that the participant was last known to be alive or the date of study cutoff, whichever came first. OS and the corresponding 2-sided 95% CI was analyzed using the Kaplan-Meier method.
Time Frame: From date of first dose of study drug until date of death from any cause or up to data cutoff (31 May 2013), up to approximately 3.25 years
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eribulin Mesylate Plus Erlotinib, 21 Day Regimen | Eribulin Mesylate Plus Erlotinib, 28 Day Regimen
Number analyzed (Participants) | 63 | 60
Months | 7.6 [6.3 to 11.0] | 8.5 [6.2 to 13.1]

ADVERSE EVENTS:
Time Frame: From date of administration of first dose up to 30 days after the last dose, or up to approximately 6 years 11 months
Description: Treatment-emergent adverse events (TEAEs) included adverse events that occurred from the first dose of study drug to 30 days after the last dose of study drug, or that were present prior to the first dose of study drug administration but worsened in severity during the study.
Arm/Group | Eribulin Mesylate, 21 Day Cycle | Eribulin Mesylate, 28 Day Cycle
All-Cause Mortality (participants affected / at risk) | 59/63 | 51/60
Serious Adverse Events (participants affected / at risk) | 38/63 | 27/60
Other Adverse Events (participants affected / at risk) | 61/63 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate, 21 Day Cycle (N=63) | Eribulin Mesylate, 28 Day Cycle (N=60)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 2
Neutropenia (Blood and lymphatic system disorders) | 4 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 1
Asthenia + Fatigue (General disorders) | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Haematoma infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 4 | 3
Sepsis (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 4 | 3
White blood cell count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cataract (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate, 21 Day Cycle (N=63) | Eribulin Mesylate, 28 Day Cycle (N=60)
Anaemia (Blood and lymphatic system disorders) | 19 | 25
Leukopenia (Blood and lymphatic system disorders) | 5 | 8
Neutropenia (Blood and lymphatic system disorders) | 29 | 25
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 3
Tachycardia (Cardiac disorders) | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 13 | 21
Diarrhoea (Gastrointestinal disorders) | 34 | 26
Dyspepsia (Gastrointestinal disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 20 | 23
Stomatitis (Gastrointestinal disorders) | 21 | 11
Vomiting (Gastrointestinal disorders) | 14 | 16
Asthenia (General disorders) | 5 | 6
Asthenia + Fatigue (General disorders) | 31 | 33
Chills (General disorders) | 5 | 2
Fatigue (General disorders) | 29 | 30
Mucosal inflammation (General disorders) | 8 | 1
Oedema peripheral (General disorders) | 5 | 5
Pyrexia (General disorders) | 12 | 5
Pneumonia (Infections and infestations) | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 8 | 7
Urinary tract infection (Infections and infestations) | 6 | 3
Neutrophil count decreased (Investigations) | 8 | 9
Weight decreased (Investigations) | 7 | 6
White blood cell count decreased (Investigations) | 6 | 7
Decreased appetite (Metabolism and nutrition disorders) | 18 | 24
Dehydration (Metabolism and nutrition disorders) | 3 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 16 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Arthralgia + Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Acne (Skin and subcutaneous tissue disorders) | 3 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 20 | 12
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 10 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 8
Rash (Skin and subcutaneous tissue disorders) | 28 | 15
Dizziness (Nervous system disorders) | 6 | 9
Dysgeusia (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 10 | 7
Peripheral Neuropathy (Nervous system disorders) | 5 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 6
Insomnia (Psychiatric disorders) | 4 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 14
Dry mouth (Gastrointestinal disorders) | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 1
Malaise (General disorders) | 2 | 3
Pain (General disorders) | 1 | 3
Bronchitis (Infections and infestations) | 3 | 3
Nasopharyngitis (Infections and infestations) | 0 | 3
Oral candidiasis (Infections and infestations) | 2 | 3
Paronychia (Infections and infestations) | 4 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 5
Blood phosphorus decreased (Investigations) | 0 | 3
Breath sounds abnormal (Investigations) | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Neuropathy based on broad MedDRA SMQ (Musculoskeletal and connective tissue disorders) | 4 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Hypoaesthesia (Nervous system disorders) | 3 | 3
Neuropathy based on broad MedDRA SMQ (Nervous system disorders) | 8 | 12
Neuropathy peripheral (Nervous system disorders) | 2 | 4
Anxiety (Psychiatric disorders) | 4 | 2
Renal failure (Renal and urinary disorders) | 0 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3
Hypotension (Vascular disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other